CLINICAL TRIAL: NCT02595034
Title: A Randomized Double Blind Multiple Center Placebo Controlled Study Comparing CLBG and Benzoyl Peroxide Gel 1%/5% to BenzaClin® (Clindamycin 1%/Benzoyl Peroxide 5%) Topical Gel in the Treatment of Acne Vulgaris
Brief Title: A Study CLBG and Benzoyl Peroxide Gel 1%/5% to BenzaClin® Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBG 1412
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clindamycin/BP Gel 1%5% (Experimental): Clindamycin and Benzoyl Peroxide Gel 1%/5% applied twice daily (morning and evening) for 70 days (10 weeks).
  Interventions: Drug: Clindamycin and Benzoyl Peroxide Gel 1%5%
- BenzaClin® Topical Gel (Active Comparator): BenzaClin® (clindamycin 1%/benzoyl peroxide 5%) Topical Gel applied twice daily (morning and evening) for 70 days (10 weeks).
  Interventions: Drug: BenzaClin® Topical Gel
- Placebo (Placebo Comparator): Placebo (vehicle of the test product) applied twice daily (morning and evening) for 70 days (10 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin and Benzoyl Peroxide Gel 1%5% — Clindamycin and Benzoyl Peroxide Gel 1%5% (Taro Pharmaceuticals Inc.)
  Other Names: Active
  Arms: Clindamycin/BP Gel 1%5%
Drug: BenzaClin® Topical Gel — BenzaClin® (clindamycin 1%/benzoyl peroxide 5%) Topical Gel (Sanofi Aventis, U.S.)
  Other Names: Active
  Arms: BenzaClin® Topical Gel
Drug: Placebo — Placebo (vehicle of the test product) (Taro Pharmaceuticals Inc.)
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
This study is to evaluate the therapeutic equivalence and safety of Clindamycin and Benzoyl Peroxide Gel 1%/5% and BenzaClin® (clindamycin 1%/benzoyl peroxide 5%) Topical Gel

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the therapeutic equivalence and safety of Clindamycin and Benzoyl Peroxide Gel 1%/5% (Taro Pharmaceuticals Inc.) and BenzaClin® (clindamycin 1%/benzoyl peroxide 5%) Topical Gel (Sanofi Aventis, US) in the treatment of acne vulgaris and to demonstrate the superiority of the efficacy of the test and reference products over the placebo control

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or nonpregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
2. On the face, ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤ 2 nodulocystic lesions (i.e., nodules and cysts).
3. Investigator's Global Assessment (IGA) of acne severity grade 2, 3, or 4
4. Willing to refrain from use of all other topical acne medications or antibiotics during the 10week treatment period.
5. If female of childbearing potential, willing to use an acceptable form of birth control during the study.

Exclusion Criteria

1. Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
2. Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.
3. History of hypersensitivity or allergy to benzoyl peroxide or clindamycin and/or any of the study medication ingredients.
4. Use within 6 months prior to baseline of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
5. Use for less than 3 months prior to baseline of estrogens or oral contraceptives; use of such therapy must remain constant throughout the study.
6. Use on the face within 1 month prior to baseline or during the study of: 1) cryodestruction or chemodestruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy.
7. Use within 1 month prior to baseline of: 1) spironolactone, 2) systemic steroids, 3) systemic antibiotics, 4) systemic treatment for acne vulgaris (other than oral retinoids, which require a 6-month washout), or 5) systemic anti-inflammatory agents.
8. Use within 2 weeks prior to baseline of: 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti-inflammatory agents, 5) medicated cleansers or 6) topical antibiotics.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count | Week 10 (day 70)
  Mean percent change from baseline to week 10 (study day 70) in the inflammatory (papules and pustules) lesion counts.
Change in non-inflammatory lesion count | Week 10 (day 70)
  Mean percent change from baseline to week 10 (study day 70) in the non-inflammatory (open and closed comedones) lesion counts.

SECONDARY OUTCOMES:
Clinical response of success | Week 10 (day 70)
  The proportion of subjects with a clinical response of success at week 10 (study day 70) defined as an Investigator's Global Assessment score at least 2 grades less than baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No